CLINICAL TRIAL: NCT01600924
Title: Study on the Assessment of Determinants of Muscle and Bone Strength Abnormalities in Diabetes
Acronym: SAMBA
Status: Active, not recruiting | Type: Observational
Sponsor: Metabolic Fitness Association, Italy (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giuseppe Pugliese, MD, PhD, Metabolic Fitness Association, Italy
Other Study IDs: MFA-12-02
Record Dates: First submitted 2012-05-16; First posted 2012-05-17 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: diabetes mellitus; muscle strength; bone strength; cardiovascular risk factors; diabetic complications
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus; Diabetes Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, plasma, serum and urine samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This project will assess the independent predictors of impaired muscle and bone strength through a longitudinal observation of a cohort of subjects with type 1 and 2 diabetes consecutively attending an outpatients diabetes clinics for the annual screening of complications.

DETAILED DESCRIPTION:
Impaired muscle strength has been reported in subjects with type 1 and type 2 diabetes as a late complication of severe diabetic peripheral neuropathy (DPN). However, reduction of muscle strength has been shown to occur earlier in the course of diabetes, independent of DPN. Individuals with diabetes also show an increased risk of bone fractures, which seems to be dependent on mechanisms at least partly differing from those associated with senile or post-menopausal osteoporosis. Interestingly, bone mineral density (BMD) was found to be reduced in patients with type 1 diabetes in most but not all studies, whereas cross-sectional surveys in subjects with type 2 diabetes reported normal or even increased BMD, despite the overall increase in fracture risk, thus suggesting reduced bone quality.

This project will assess the independent predictors of impaired muscle and bone strength in subjects with type 1 and 2 diabetes. This is a longitudinal observational study enrolling 500 consecutive patients who have attended an outpatients diabetes clinics since 2008 for the annual screening of complications and followed-up for at least 4 years.

Isometric upper and lower body muscle strength will be assessed by dynamometry, whereas bone strength will be evaluated by qualitative ultrasound (QUS).

The following information will be collected by a structured interview: demographics, alcohol intake, smoking status, known diabetes duration, current treatment including glucose, blood pressure (BP) and lipid-lowering, anti-platelet and anti-coagulant therapy, with indication of the class of drug, previous documented retinal photocoagulation or major acute CVD events, including myocardial infarction, stroke, foot ulcer or gangrene, amputation, coronary, carotid, and lower limb revascularization. Physical activity (PA) level will be assessed by the use of the Minnesota Leisure Time PA (LTPA) questionnaire.

Maximal oxygen consumption (Vo2max) will be assessed at the treadmill, using a modified Balke and Ware protocol, with direct measurement of oxygen consumption using the gas exchange analyzer (FitMate, Cosmed, Rome, Italy). Body weight and height will be measured with scale and stadiometer, and body mass index (BMI) will be then calculated. Waist circumference will be measured as the minimum circumference between the lower rib margin and the iliac crest while. Fat mass and fat free mass will be assessed using a whole body densitometer (QDR 2000plus, Hologic Italy, Rome, Italy). BP will be measured with a mercury sphygmomanometer on the right arm after the patient has been seated for at least 5 min. Ankle-brachial index (ABI) will be assessed by measuring systolic BP at the ankle and brachial level using a mercury sphygmomanometer and a handheld continuous wave Doppler device (Super Doppler 2, Huntleight Healthcare, MedicalResources.com, Lewis Center, OH). Carotid intima-media thickness (IMT) will be assessed by color-coded duplex sonography (Agilent HP ImagePoint HX, Hewlett Packard, USA). Diabetic retinopathy (DR) will be evaluated by fundus examination in mydriasis. The distal latencies, amplitudes, and nerve conduction velocities of the peroneal motor and sural sensory nerves will be measured bilaterally, using a Medelec MS 928 Neurostar (Oxford Instruments Medical, Old Woking,U.K.), together with the vibration perception threshold (VPT) in the left and right malleolus and hallux by the use of Biothesiometer (Horwell, Nottingham, U.K.). Autonomic function will be assessed by cardiovascular autonomic reflex tests (CARTs), HR response to deep breathing (expiration-to-inspiration [EI] ratio), cough test (CT ratio), and standing, (30:15 ratio) and systolic BP response to standing (systolic - diastolic BP).

HbA1c will be assessed by a DCCT-aligned high-performance liquid chromatography method (Adams TMA1C HA-8160, Menarini Diagnostics, Florence, Italy). Fasting and post-prandial (1 hour after a standard breakfast) glucose, triglycerides, total and HDL cholesterol, nitrogen, and uric acid will be measured by standard analytical methods using the VITROS 5,1 FS Chemistry System (Ortho-Clinical Diagnostics, Inc, Raritan, NJ, USA) and LDL cholesterol will be calculated by the Friedwald formula. Serum creatinine will be measured by the modified Jaffe method and estimated glomerular filtration rate (eGFR) will be calculated by the four-variable Modification of Diet in Renal Disease (MDRD) Study or the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation. Albuminuria will be assessed as albumin/creatinine ratio by measuring albumin and creatinine concentration by immunonephelometry and the modified Jaffe method, respectively, in early-morning, first-voided urine samples. Subjects will be then classified as having no CKD or CKD stages 1-5, based on the value of eGFR and the presence or absence of micro or macroalbuminuria, according to the NKF's Kidney Disease Outcomes Quality Initiative (KDOQI).

The role of cardiovascular risk factors and complications at baseline as independent predictors of reduced muscle and bone strength will be assessed (primary endpoints), together with relation of changes over time in these factors with impairment of muscle and bone strength (secondary endpoints).

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 or 2 diabetes

Exclusion Criteria:

* Patients with any condition precluding mobility

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients clinics
Sampling Method: Probability Sample
Enrollment: 1018 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Independent predictors of reduced muscle and bone strength | 4 years
  Baseline parameters predicting reduction of muscle and bone strength

SECONDARY OUTCOMES:
Relation of changes in predictors with reduced muscle and bone strength | 4 years
  Relation of changes over time in predictors with reduced muscle and bone strength

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Balducci, MD, Study Director — Sant'Andrea Hospital, Diabetes Unit
Locations (1):
- University of Rome La Sapienza, Department of Clinical and Molecular Medicine, Sant'Andrea Hospital, Diabetes Unit, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andreassen CS, Jakobsen J, Andersen H. Muscle weakness: a progressive late complication in diabetic distal symmetric polyneuropathy. Diabetes. 2006 Mar;55(3):806-12. doi: 10.2337/diabetes.55.03.06.db05-1237. PMID 16505247
- [Background] Andreassen CS, Jakobsen J, Ringgaard S, Ejskjaer N, Andersen H. Accelerated atrophy of lower leg and foot muscles--a follow-up study of long-term diabetic polyneuropathy using magnetic resonance imaging (MRI). Diabetologia. 2009 Jun;52(6):1182-91. doi: 10.1007/s00125-009-1320-0. Epub 2009 Mar 12. PMID 19280173
- [Background] Stenholm S, Harkanen T, Sainio P, Heliovaara M, Koskinen S. Long-term changes in handgrip strength in men and women--accounting the effect of right censoring due to death. J Gerontol A Biol Sci Med Sci. 2012 Oct;67(10):1068-74. doi: 10.1093/gerona/gls064. Epub 2012 Mar 15. PMID 22421705
- [Background] IJzerman TH, Schaper NC, Melai T, Meijer K, Willems PJ, Savelberg HH. Lower extremity muscle strength is reduced in people with type 2 diabetes, with and without polyneuropathy, and is associated with impaired mobility and reduced quality of life. Diabetes Res Clin Pract. 2012 Mar;95(3):345-51. doi: 10.1016/j.diabres.2011.10.026. Epub 2011 Nov 21. PMID 22104262
- [Background] Vestergaard P. Discrepancies in bone mineral density and fracture risk in patients with type 1 and type 2 diabetes--a meta-analysis. Osteoporos Int. 2007 Apr;18(4):427-44. doi: 10.1007/s00198-006-0253-4. Epub 2006 Oct 27. PMID 17068657
- [Background] Merlotti D, Gennari L, Dotta F, Lauro D, Nuti R. Mechanisms of impaired bone strength in type 1 and 2 diabetes. Nutr Metab Cardiovasc Dis. 2010 Nov;20(9):683-90. doi: 10.1016/j.numecd.2010.07.008. PMID 20934862
- [Background] Melton LJ 3rd, Leibson CL, Achenbach SJ, Therneau TM, Khosla S. Fracture risk in type 2 diabetes: update of a population-based study. J Bone Miner Res. 2008 Aug;23(8):1334-42. doi: 10.1359/jbmr.080323. PMID 18348689
- [Background] Howe TE, Shea B, Dawson LJ, Downie F, Murray A, Ross C, Harbour RT, Caldwell LM, Creed G. Exercise for preventing and treating osteoporosis in postmenopausal women. Cochrane Database Syst Rev. 2011 Jul 6;2011(7):CD000333. doi: 10.1002/14651858.CD000333.pub2. PMID 21735380
- [Derived] Conti F, Balducci S, Pugliese L, D'Errico V, Vitale M, Alessi E, Salerno G, Iacobini C, Menini S, Bollanti L, Nicolucci A, Pugliese G. Correlates of Calcaneal Quantitative Ultrasound Parameters in Patients with Diabetes: The Study on the Assessment of Determinants of Muscle and Bone Strength Abnormalities in Diabetes. J Diabetes Res. 2017;2017:4749619. doi: 10.1155/2017/4749619. Epub 2017 Sep 19. PMID 29057273
- [Derived] Balducci S, Sacchetti M, Orlando G, Salvi L, Pugliese L, Salerno G, D'Errico V, Iacobini C, Conti FG, Zanuso S, Nicolucci A, Pugliese G; Study on the Assessment of Determinants of Muscle and Bone Strength Abnormalities in Diabetes SAMBA Investigators. Correlates of muscle strength in diabetes: The study on the assessment of determinants of muscle and bone strength abnormalities in diabetes (SAMBA). Nutr Metab Cardiovasc Dis. 2014 Jan;24(1):18-26. doi: 10.1016/j.numecd.2013.04.010. Epub 2013 Oct 3. PMID 24095149
- See also: Study protocol — http://www.metabolicfitness.it/